CLINICAL TRIAL: NCT01804712
Title: A Pilot Study of Rituximab Neoadjuvant Therapy in Patients With High Risk Prostate Cancer Scheduled to Undergo Radical Prostatectomy
Brief Title: Rituximab Neoadjuvant Therapy in Patients With Prostate Cancer Scheduled to Undergo Radical Prostatectomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stephen Howell, M.D. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Stephen Howell, M.D., Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121451
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Castration-resistant; Rituximab; neoadjuvant; Rituxan
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab (Experimental): Rituximab will be administered intravenously at a dose of 375 mg/m2 of body surface area once per week for 4 weeks (Days 1, 8, 15, and 22 of a 28-day cycle).
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — Rituximab will be administered intravenously at a dose of 375 mg/m2 of body surface area once per week for 4 weeks (Days 1, 8, 15, and 22 of a 28-day cycle).
  Other Names: Rituxan

SUMMARY:
There is now substantial evidence that B cells are recruited into prostate cancers by CXCL13 released by the tumor cells. B cells release lymphotoxin which drives malignant cell proliferation through the NFkB pathway. This is a pilot trial in 18 patients to determine whether depletion of B cells by rituximab will result in a decrease in the extent of B cell infiltration of the prostatic cancer. The extent of infiltration in the diagnostic biopsy will be compared to that in the prostatectomy samples following administration of 4 weekly doses of rituximab.

DETAILED DESCRIPTION:
This is an open label, single institution, pilot study of rituximab neoadjuvant therapy in patients with high risk prostate cancer scheduled to undergo radical prostatectomy. Prior to prostatectomy, patients will receive one treatment cycle (28 days) of rituximab 375 mg/m2 intravenously once weekly. Patients will be scheduled to undergo radical prostatectomy within two weeks of completing study treatment. Tissue from prostatectomy will be used for immunohistochemistry (IHC) staining of pharmacodynamic markers.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide written informed consent.
* Patient has EITHER:

  * A Kattan nomogram predicted probability of being disease free 5 years after surgery of < 60%, OR
  * A Gleason sum ≥ 8.
* Indicated for radical prostatectomy.

Note: candidates for radical prostatectomy are still eligible even if they have a history of deep venous thrombosis, pulmonary embolism, and/or cerebrovascular accident or currently requiring systemic anticoagulation.

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Appendix A).
* Males aged ≥ 18 years.
* Adequate organ function as defined below measured within 21 days of study entry:
* Hematology:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin ≥ 9.0 g/dL
  * White blood cell (WBC) count ≥ 3.0 x 109/L
* Biochemistry:

  * Aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/SGOT) and alanine transaminase/serum glutamate pyruvate transaminase (ALT/SGPT) ≤ 2 x institution's upper limit of normal (ULN)
  * Total bilirubin <1.5 times ULN
  * Serum creatinine and blood urea nitrogen (BUN)<1.5 times ULN
  * Na, K Cl, carbon dioxide (CO2), Ca, phosphate (PO4) within institutional limits
* Available prostate biopsy specimen which is evaluable for B lymphocyte count.

Exclusion Criteria:

* Received prior treatment for prostatic adenocarcinoma including prior surgery (excluding TURP), radiation therapy, or chemotherapy.
* Current or past use of investigational agents within 4 weeks of study enrollment.
* Evidence of metastatic disease on cross sectional imaging or bone scan.
* History of hepatitis B or C, hepatitis immunodeficiency virus (HIV), tuberculosis or a chronic infection of any type.
* Positive test results for chronic hepatitis B infection (defined as positive HBsAg serology).
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Histologic response rate after one cycle of rituximab | 1 treatment cycle (28 days)

SECONDARY OUTCOMES:
Change in prostate-specific antigen (PSA) | from Day 1 to Day 29
Change in peripheral blood B cell number | from Day 1 to Day 29
Change in serum CXCL13 level | from Day 1 to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Howell, MD, Principal Investigator — University of California Medical Center
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

REFERENCES:
- [Derived] Ryan ST, Zhang J, Burner DN, Liss M, Pittman E, Muldong M, Shabaik A, Woo J, Basler N, Cunha J, Shalapour S, Estrada MV, Karin M, Messer K, Howell S, Kane CJ, Jamieson CAM. Neoadjuvant rituximab modulates the tumor immune environment in patients with high risk prostate cancer. J Transl Med. 2020 May 28;18(1):214. doi: 10.1186/s12967-020-02370-4. PMID 32466781